CLINICAL TRIAL: NCT05409664
Title: Peer Coaching for Physical Activity Promotion Among Breast Cancer Survivors: Adapting an Efficacious Intervention to Prepare for Implementation
Brief Title: Moving Forward Together 4
Acronym: MFT4
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: University of Colorado, Denver (Other); Brown University (Other); InquisitHealth, Inc. (Other)
Responsible Party: Principal Investigator, Bernardine Pinto, Associate Dean for Research, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00117242
Record Dates: First submitted 2022-05-12; First posted 2022-06-08 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Physical Inactivity
Keywords: Peer support
MeSH Terms: conditions — Breast Neoplasms; Sedentary Behavior | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial. Participants will be randomly assigned to a intervention group or a control group. The study duration will be 3-months for both groups; assessments will be completed pre- and post-intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- webMFT (Experimental): Survivors randomized to webMFT will receive the evidence-based intervention for moderate-to-vigorous physical activity (MVPA) promotion that consists of MVPA counseling matched to patients' motivational readiness, and self-monitoring of MVPA (via Fitbit Inspire 2). The goal for the 3-month program will be to gradually increase the amount of moderate-intensity aerobic exercise that is performed, to the current national recommendations of at least 150 minutes of MPVA per week. Our goal is to promote aerobic exercise that is safe and enjoyable, such as walking.
  Interventions: Behavioral: Physical activity adoption
- MVPA tracking (Active Comparator): These survivors will be asked to self-monitor moderate-to-vigorous physical activity (MVPA) participation by wearing the Fitbit Inspire 2 each day over 12 weeks. This group will not receive the MVPA counseling from the coaches.
  Interventions: Behavioral: Self monitoring

INTERVENTIONS:
Behavioral: Physical activity adoption — webMFT will be delivered via a web-based platform. Coaches will be trained to deliver the intervention prior to being assigned a study participant. Upon successful completion of the informed consent for coaches and participants, coaches will be assigned a participant for their 3-month duration in the study. Coaches and participants will complete weekly phone calls focused on increasing the participants' MVPA up to the recommended 150 min/week.
  Arms: webMFT
Behavioral: Self monitoring — Participants will be asked to gradually increase their activity up to the recommended 150 minutes of moderate-intensity/week during the 12-week intervention. Self-monitoring will be completed using a Fitbit tracker.
  Arms: MVPA tracking

SUMMARY:
This is a 3-month physical activity intervention aimed to increase moderate-intensity activity among previously inactive breast cancer survivors. Participants will be eligible if they are not currently active, and have recently been diagnosed with breast cancer. Upon eligibility, participants will be randomized into one of two groups. The intervention group will receive weekly guidance from a peer coach to increase their activity throughout the three month intervention. The control group will be encouraged to self-monitor their physical activity throughout the three month intervention. Both groups will receive a Fitbit. Peer coaches will be trained to deliver the physical activity program using a web-based platform; all calls will be virtual. Participants will be assessed before and after the intervention.

ELIGIBILITY:
Participants:

Inclusion Criteria:

* Diagnosed in the past 5 years with Stage 0-3 breast cancer
* Able to read and speak English
* Ambulatory
* Sedentary (<30 minutes of vigorous-intensity physical activity, <90 min of moderate-intensity physical activity in the past 6 months)
* Able to walk unassisted
* Access to a smartphone with Bluetooth and internet

Exclusion Criteria:

* Stage 4 cancer
* Medical or psychiatric problem that may interfere with protocol adherence

Peer Mentor Coaches:

Inclusion criteria:

* Current peer coach (at least one year)
* Have a valid email address, telephone access, and access to a tablet/computer
* Willing to participate in group training
* Willing to be supervised using platform
* Currently exercise for at least 60 min/week of moderate-intensity activity

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Accelerometer measured moderate-to-vigorous activity | 3-month intervention
  Minutes of moderate-to-vigorous intensity activity at 3-month follow-up

SECONDARY OUTCOMES:
Self-Reported Quality of Life | Pre-intervention and post 3-month intervention
  Assessed via FACT-B, validated questionnaire
Self-Reported Physical Functioning | Pre-intervention and post 3-month intervention
  Assessed via SF-36, validated questionnaire
Self-Reported Mood | Pre-intervention and post 3-month intervention
  Assessed via Profile of Mood States, validated questionnaire
Self-Reported Fatigue | Pre-intervention and post 3-month intervention
  Assessed via FACIT-F, validated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bernardine M. Pinto, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared upon request.

REFERENCES:
- [Derived] Ostendorf DM, Huebschmann AG, Wickersham KE, Kindred M, Pinto BM. Adopting and implementing an efficacious peer-delivered physical activity program for web platform delivery in survivors of breast cancer: organizational readiness and perspectives. Transl Behav Med. 2025 Jan 16;15(1):ibaf051. doi: 10.1093/tbm/ibaf051. PMID 41005365
- [Derived] Pinto BM, Kindred M, Dunsiger S, Mitchell S, Patel A, Ostendorf D, Huebschmann AG. Effects of web platform delivery of a physical activity program for breast cancer survivors: a randomized controlled trial. J Cancer Surviv. 2025 May 27. doi: 10.1007/s11764-025-01811-7. Online ahead of print. PMID 40423894
- [Derived] Pinto BM, Patel A, Ostendorf DM, Huebschmann AG, Dunsiger SI, Kindred MM. Adapting an Efficacious Peer-Delivered Physical Activity Program for Survivors of Breast Cancer for Web Platform Delivery: Protocol for a 2-Phase Study. JMIR Res Protoc. 2024 Jun 19;13:e52494. doi: 10.2196/52494. PMID 38896452